CLINICAL TRIAL: NCT01985373
Title: Pharmacokinetics and Safety of the Intravenous Human Immunoglobulin Product Nanogam 100 mg/ml
Brief Title: Pharmacokinetics and Safety of IVIG Nanogam 100 mg/ml
Acronym: Nanogam
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD2012.02; 2012-005727-32 (EudraCT Number)
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Primary Immunodeficiency
Keywords: intravenous immunoglobulin; pharmacokinetics; 10% IVIG
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous immunoglobulin infusion (Experimental): One intravenous infusion with Nanogam 50 mg/ml and 4 with Nanogam 100 mg/ml (0.2-0.8 g/kg)
  Interventions: Drug: Intravenous immunoglobulin infusion

INTERVENTIONS:
Drug: Intravenous immunoglobulin infusion — Blood samples are drawn before infusion with Nanogam 50 and Nanogam 100 mg/ml and IgG levels are determined to study PK
  Other Names: Nanogam

SUMMARY:
Intravenous immunoglobulin (IVIG) is used for treatment of a heterogeneous group of immune related disorders both as immune-replacement and immune-modulating therapy. Sanquin developed a 100 mg/ml IVIg product (Nanogam 100 mg/ml). Patient will receive one infusion with Nanogam 50 mg/ml as they used to (same dose) and subsequently 4 infusions with Nanogam 100 mg/ml (same dose). Aim is to show bioequivalency between the 50 mg/ml and the 100 mg/ml product of Sanquin.

ELIGIBILITY:
Inclusion Criteria:

* Primary a- or hypogammaglobulinemia, particularly patients with XLA or CVID
* Stabilised on treatment with Nanogam 50 mg/ml with 2-4 weeks intervals in an hospital or at home and willing to be treated with 1 infusion of Nanogam 50 mg/ml and 4 infusions of Nanogam 100 mg/ml at the hospital
* A stable clinical situation (no activity of any other disease; a stable immunoglobulin dose and frequency)
* Age >= 18 years
* The patient has signed the consent form

Exclusion Criteria:

* Known with allergic reactions against human plasma or plasma products
* Having an ongoing progressive disease, including HIV infection
* Pregnancy or lactation
* Known with insufficiency of coronary or cerebral circulation
* Having renal insufficiency (plasma creatinin > 115µmol/L)
* Having IgA deficiency and anti-IgA antibodies have been detected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
IgG trough levels | before infusion
  Comparison IVIG 5% and 10%
plasma concentration-time curve | predose, 1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days post-dose
  Comparison IVIG 5% and 10%
half-life | predose, 1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days post-dose
  Comparison IVIG 5% and 10%
area under the curve | predose, 1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days post-dose
  Comparison IVIG 5% and 10%
volume of distribution | predose, 1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days post-dose
  Comparison IVIG 5% and 10%
Cmax | predose, 1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days post-dose
  Comparison IVIG 5% and 10%
Tmax | predose, 1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days post-dose
  Comparison IVIG 5% and 10%
elimination rate constant(s) | predose, 1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days post-dose
  Comparison IVIG 5% and 10%

SECONDARY OUTCOMES:
Adverse Events | from first till 3 weeks after last infusion (11-19 weeks dependent on infusion frequency)
  number and type

CONTACTS AND LOCATIONS:
Overall Officials: F P Kroon, PhD, MD, Principal Investigator — LUMC
Locations (4):
- Netherlands (4):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - UMCG, Groningen
  - LUMC, Leiden
  - UMC St. Radboud, Nijmegen